CLINICAL TRIAL: NCT01642225
Title: Desensitization Protocol for Deceased Donor List
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Junichiro Sageshima, Associate Professor of Clinical, University of Miami
Other Study IDs: 20120052
Record Dates: First submitted 2012-07-12; First posted 2012-07-17 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Transplant; Failure, Kidney

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Purpose of the study:

The specific aims of this study are to evaluate overall efficacy and safety of the pre-transplant IVIG treatment in our transplant center since 2007 and to identify factors affecting treatment outcomes in order to improve patient selection and treatment protocols for future patients.

DETAILED DESCRIPTION:
Background:

Intravenous immunoglobulin (IVIG) infusion is one of several novel approaches to decrease antibody levels for highly sensitized kidney transplant candidates [1, 2]. This approach can potentially give a chance of kidney transplantation to end-stage renal failure patients who could never receive transplantation because of high levels of antibodies and persistent positive crossmatches to all potential kidney donors. Many transplant centers have used this strategy in order to increase transplant rates of highly sensitized patients with various levels of anti-HLA antibodies. However, the responses to the treatment seem to be different in each patient and factors affecting treatment outcome have yet to be determined.

ELIGIBILITY:
Inclusion Criteria:

* Recent (< 3 months) high levels of anti-HLA antibodies (at least one cPRA ≥ 40%).
* Waiting time greater than 1 year for blood type AB, 2 years for blood types A, B, or O.

Exclusion Criteria:

* Female subject is pregnant or lactating.
* Subject has an uncontrolled concomitant infection or any other unstable medical condition (e.g., uncontrolled cardiovascular disease) that could interfere with the study objectives.
* Subject has an uncontrolled active hepatitis B, hepatitis C, or HIV infection.
* Subject has a current malignancy or a recent history of any malignancy that is deemed to be contraindicated to kidney transplantation.
* Subject has a psychiatric illness that, in the judgment of caring physicians, may interfere with study participation.

Ages: 7 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 100 subjects are expected to participate from 2007 to current, and another 100 subjects are expected to participate during the next 12-month period.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Anti HLA antibody level | after IVIG infusion

SECONDARY OUTCOMES:
Number of patients transplanted | at the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Junichiro Sageshima, M.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States